CLINICAL TRIAL: NCT06582030
Title: Stop Addiction Stigma Training Workshop With Case Vignettes to Decrease Stigmatizing Attitudes Toward People With Substance Abuse Disorders
Brief Title: Stop Addiction Stigma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Gretchen A McNally, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: OSU-23194; NCI-2024-04797 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-06-27; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Restraint, Physical; Outcome Assessment, Health Care; Observational Studies as Topic; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Group A (chronically relapsing brain disease vignette, SAS) (Experimental): Participants view the chronically relapsing brain disease vignette and attend a SAS workshop on study.
  Interventions: Behavioral: Assessment; Other: Educational Activity
- Group B (brain disease vignette, SAS) (Experimental): Participants view the brain disease vignette and attend a SAS workshop on study.
  Interventions: Behavioral: Assessment; Other: Educational Activity; Other: Training
- Group C (disease vignette, SAS) (Experimental): Participants view the disease vignette and attend a SAS workshop on study.
  Interventions: Behavioral: Assessment; Other: Educational Activity; Other: Training
- Group D (illness vignette, SAS) (Experimental): Participants view the illness vignette and attend a SAS workshop on study.
  Interventions: Behavioral: Assessment; Other: Educational Activity; Other: Training
- Group E (disorder vignette, SAS) (Experimental): Participants view the disorder vignette and attend a SAS workshop on study.
  Interventions: Behavioral: Assessment; Other: Educational Activity; Other: Training
- Group F (problem vignette, SAS) (Experimental): Participants view the problem vignette and attend a SAS workshop on study.
  Interventions: Behavioral: Assessment; Other: Educational Activity; Other: Training

INTERVENTIONS:
Behavioral: Assessment — Ancillary studies
  Other Names: Assess; Study Assessment; Study Observation
Other: Educational Activity — View the chronically relapsing brain disease vignette
  Arms: Group A (chronically relapsing brain disease vignette, SAS)
Other: Educational Activity — View the brain disease vignette
  Arms: Group B (brain disease vignette, SAS)
Other: Educational Activity — View the disease vignette
  Arms: Group C (disease vignette, SAS)
Other: Educational Activity — View the illness vignette
  Arms: Group D (illness vignette, SAS)
Other: Educational Activity — View the disorder vignette
  Arms: Group E (disorder vignette, SAS)
Other: Educational Activity — View the problem vignette
  Arms: Group F (problem vignette, SAS)
Other: Training — Attend a SAS workshop
  Other Names: Training Programs
  Arms: Group B (brain disease vignette, SAS); Group C (disease vignette, SAS); Group D (illness vignette, SAS); Group E (disorder vignette, SAS); Group F (problem vignette, SAS)

SUMMARY:
This clinical trial evaluates the impact of a Stop Addiction Stigma (SAS) training workshop with a short description of the conditions related to addiction (vignettes) on stigmatizing attitudes toward individuals with substance abuse disorders. Reviews have shown that patients with substance abuse disorders have experienced negative attitudes from their health care providers. Negative attitudes may lead to less involvement from the provider and the patient and may lead to less effective care. Using case vignettes with a SAS workshop may be an effective method to help people learn about addiction, reduce the stigma toward addiction and improve the quality of health care.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To describe the impact of SAS training on participants' responses to people with a substance impairment.

SECONDARY OBJECTIVES:

I. To evaluate the feasibility of stigma training workshops on stigmatizing attitudes health care personnel.

II. To explore the maintainability of responses over time. III. To explore relationships between language and stigmatizing attitudes.

OUTLINE: Participants are randomized to 1 of 6 group case vignettes.

GROUP A (CHRONICALLY RELAPSING BRAIN DISEASE): Participants view the chronically relapsing brain disease vignette and attend a SAS workshop on study.

GROUP B (BRAIN DISEASE): Participants view the brain disease vignette and attend a SAS workshop on study.

GROUP C (DISEASE): Participants view the disease vignette and attend a SAS workshop on study.

GROUP D (ILLNESS): Participants view the illness vignette and attend a SAS workshop on study.

GROUP E (DISORDER): Participants view the disorder vignette and attend a SAS workshop on study.

GROUP F (PROBLEM): Participants view the problem vignette and attend a SAS workshop on study.

ELIGIBILITY:
Inclusion Criteria:

* Employee of Ohio State University Wexner Medical Center (OSUWMC)
* Age ≥ 18 years
* Participants must be able to read and comprehend survey items

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Stigmatizing attitudes | Before, immediately after and 8 weeks after the session
  Stigmatizing attitudes will be measured with the Stigma and Attribution Assessment. The assessment score will be compared both between and within participants for each case vignette. Results will be reported with descriptive statistics, including means and standard deviations or medians and first-third quartiles for continuous variables, and frequencies and percentages for discrete variables.The linear mixed effect model will be used to study the repeated stigma and attribution measures over time (pre-workshop, immediately post-workshop, and 8 weeks post-workshop) within 6 vignettes as well as the effects between the vignettes, while controlling for the potential confounding factors (e.g., sex).

SECONDARY OUTCOMES:
Attendance rate | At 90 minute session.
  The proportion of participants attending the workshop will be summarized with 95% confidence interval.
Response to post-workshop evaluations | Before, immediately following and 8 weeks after the session.
  The proportion of participants who respond to the post-workshop evaluations will be summarized with 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen A Mcnally, PhD, APRN-CNP, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

DOCUMENTS (1):
  • Informed Consent Form (2023-09-29): https://cdn.clinicaltrials.gov/large-docs/30/NCT06582030/ICF_000.pdf